CLINICAL TRIAL: NCT00406965
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of HAE1 (PRO98498) in Subjects With Moderate to Severe Allergic Asthma
Brief Title: A Study to Evaluate the Safety and Efficacy of HAE1 in Subjects With Moderate to Severe Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: HAE3973g
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Allergic Asthma

INTERVENTIONS:
Drug: HAE1 (PRO98498)

SUMMARY:
This is a Phase II, multicenter, randomized, double blind, placebo controlled, multiple-dose study designed to evaluate the efficacy, safety, and tolerability of subcutaneously administered HAE1 in subjects 12-75 years old with moderate to severe asthma whose symptoms are inadequately controlled with moderate to high-dose ICS and LABA.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form(s)
* Male and females 12-75 years of age with the diagnosis of allergic asthma for 12 months according to the standards of the American Thoracic Society
* Baseline FEV1 values ≥ 40% to ≤ 80% of the predicted normal value for the subject
* Demonstration of ≥ 12% increase in FEV1 over baseline value within 30 minutes of taking up to four puffs of albuterol (90 ug/puff)
* Treatment with ICS in doses equivalent to 250-500 ug fluticasone twice daily (BID) for 8 weeks prior to screening and as needed or regular use of bronchodilator therapy
* Treatment with a stable regimen of 50 ug salmeterol BID or 12 ug formoterol BID for at least 8 weeks prior to screening (with or without other asthma controller medications)
* A positive radioallergosorbent test (RAST) to one or more of the pertinent perennial or seasonal allergens
* Total serum IgE level ≥ 20 to ≤ 1500 IU/mL and body weight between ≥ 40 and ≤ 150 kg
* Acceptable medical history and physical examination results
* Demonstrated ability to use Mini-Wright peak flow meter for the measurement of peak expiratory flow (PEF) and a metered dose inhaler (MDI) for administration of albuterol rescue medication
* Willingness to complete the daily diary cards
* History of smoking of less than 10 pack-years and no smoking for ≥ 12 months
* For females of childbearing potential, use an effective method of contraception from screening throughout their duration of study participation (e.g., oral, mechanical, SC, or surgical contraception)
* Inadequately controlled asthma 4 weeks during the run-in period as demonstrated by either of the following: One or more nighttime awakenings per week or Asthma symptoms during the day requiring rescue medication for 2 or more days per week

Exclusion Criteria:

* Active lung disease other than asthma
* Asthma exacerbation requiring treatment with the addition of systemic (oral or IV) corticosteroids or an increase in systemic corticosteroids within 1 month prior to screening or during the run-in period
* Significant change (e.g., 50% change) in dosage of inhaled corticosteroids in daily dose or dosing schedule within 1 month of prior to the screening visit or during the run-in period
* Significant medical illness other than asthma
* Treatment with methotrexate, gold salts, cyclosporine, theophyllines, or macrolide antibiotics within 3 months prior to screening or during the run-in period
* Treatment with HAE1
* Any treatment with omalizumab
* Known hypersensitivity to the ingredients of the HAE1 formulation, to trial rescue medication (albuterol), or related drugs
* History of acute infectious sinusitis or respiratory tract infection within 1 month prior to screening or during the run-in period
* Aspirin or other nonsteroidal anti-inflammatory drug-related asthma
* Allergy vaccination therapy < 3 months of stable maintenance dose prior to screening
* Treatment with oral or parenteral corticosteroids within 1 month prior to screening or during the run-in period
* Current treatment with <beta>-blocker medications (e.g., propranolol)
* Clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening
* Abnormal chest X-ray (excluding changes consistent with asthma) within 12 months prior to screening
* Clinically significant or active systemic disease (e.g., cancer, neoplasia, infection, hematological, renal, hepatic, coronary heart disease or other cardiovascular diseases, or endocrine or gastrointestinal disease) within 3 months of screening or during the run-in period
* Inability or unwillingness to comply with study procedures and visits (e.g., spirometry, blood draws, subject diary)
* History of drug or alcohol abuse
* Elevated serum IgE levels for reasons other than allergy (e.g., parasitic infection, hyperimmunoglobulin E syndrome, Wiskott-Aldrich syndrome, or bronchopulmonary aspergillosis)
* Pregnancy or lactation
* Platelet count ≤ 110,000/mm^3 or ≤ 110 x 10^9/L at screening or the qualifying run-in visit
* Clinically significant laboratory abnormalities, which would limit participation in the study or interfere in the interpretation of study, or affect subject safety, and evaluations at screening or the qualifying run-in visit
* Treatment with an investigational drug within 1 month of screening or during the run-in period

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2006-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the change from baseline (Visit 1) in total asthma symptom score to Visit 10 (Day 140).

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and targeted adverse events and incidence of HAE-1 specific antibodies from Visit 1 to the end of the study
Change from baseline (Visit 1) in asthma symptom scores (nocturnal, morning, daytime, and total) at Visits 5, 6, 7, 8, and 10 (Days 28, 56, 84, 112, and 140)
Change from baseline (Visit 1) in the number of puffs per day of beta2-agonist rescue medication at Visits 5, 6, 7, 8, and 10 (Days 28, 56, 84, 112, and 140)
The rate of asthma exacerbations at Visit 10
Change from baseline (Visit 1) in the ACQ at Visits 5, 6, 7, 8, 10, 11, 12, 13, and 14 (Days 28, 56, 84, 112, 140, 168, 196, 224, and 252)
Change from baseline (Visit 1) in percent predicted forced expiratory volume in 1 second (FEV1) at Visits 5, 6, 7, 8, and 10 (Days 28, 56, 84, 112, and 140).

CONTACTS AND LOCATIONS:
Overall Officials: Yamo Deniz, M.D., Study Director — Genentech, Inc.